CLINICAL TRIAL: NCT05781672
Title: Longitudinal Analysis of Myocardial Function by Speckle Tracking Echocardiography and Prediction of Delayed Toxic Cardiomyopathy Associated With Anthracycline Therapy in Children
Brief Title: Prediction of Delayed Toxic Cardiomyopathy in Children
Acronym: SpeckleAnthra2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analyses will be performed with data from included patients until the end of the inclusion period. The clinical team did not wish to extend the inclusion period in order not to delay the analyses.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL22_0513
Record Dates: First submitted 2023-02-27; First posted 2023-03-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Cardiotoxicity; Childhood Cancer
Keywords: Echocardiography; Ventricular function; Stroke Volume
MeSH Terms: conditions — Cardiotoxicity; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anthra2 (Experimental): Patient will have an echocardiography with speckle tracking analysis 5 years after the end of their participation to "SpeckleAnthra" study (NCT02893787)
  Interventions: Diagnostic Test: cardiac ultrasound with speckle tracking analysis
- Control (Active Comparator): Cardiac ultrasound analysis with speckle tracking of age- and sex-matched healthy patients in the Anthra2 group
  Interventions: Diagnostic Test: cardiac ultrasound with speckle tracking analysis

INTERVENTIONS:
Diagnostic Test: cardiac ultrasound with speckle tracking analysis — Experimental group: cardiac ultrasound with speckle tracking analysis done during a regular cardiac visit planned after receiving cardiotoxic chemotherapy in childhood.
  Control group: cardiac ultrasound with speckle tracking analysis done during a cardiac visit for minor symptoms (murmur, physical aptitude).
  Advocated Tomtec software will be used to make post-processing speckle tracking analysis based on 2D ultrasound cineloop acquired during a standard echocardiography.

SUMMARY:
Longitudinal analysis of myocardial function using "Speckle Tracking Echocardiography" STE analysis and prediction of delayed toxic induced cardiomyopathy in young patients who received anthracycline therapy in childhood.

DETAILED DESCRIPTION:
Anthracycline therapy may have short-, medium- or long-term cardiac toxicity that impacts patient's life. The main recognized risk factors for delayed cardiotoxicity are cumulative anthracycline dose, female gender, association with mediastinal radiotherapy and young age at administration. Prediction of delayed cardiotoxicity in children population is still challenging.

The "Speckle Tracking Echocardiography" (STE) method, an innovative echocardiographic technique, analyses the myocardial displacement of natural acoustic markers via a software. The objective of the study is to analyze, in young patients who received anthracycline therapy in childhood, 5-years after their inclusion in the "Speckle Anthra" study and first STE results, the evolution of myocardial function using STE method.

ELIGIBILITY:
ANTHRA GROUP

Inclusion Criteria:

* Patients who were treated with anthracyclines for malignant disease between the ages of 0 and 18
* Patient aged 11 to 27 years
* Included in the "SpeckleAnthra" Study (NCT02893787)
* Discontinued chemotherapy for more than 6 years
* Patient in remission of malignant disease
* Enrolled in a social security plan
* Written informed consent from at least one legal representative for the minor patient/ Written informed consent for patients of legal age

Exclusion Criteria:

* Onset of active malignancy or recurrence of malignancy after the "Speckle Anthra" study that required resumption of chemotherapy or mediastinal radiotherapy.
* Chronic cardiac, pulmonary or muscular pathology of etiology other than secondary to anthracycline therapy
* For adult patients: subject under guardianship or curators

CONTROL GROUP

Inclusion Criteria:

* Control patient included in the "Speckle Control" study (NCT02056925)
* Had a cardiological consultation with echocardiography performed for a banal reason (heart murmur test, cardiological symptoms) and whose result was normal
* No chronic disease or long-term drug treatment

Exclusion Criteria:

* Refusal to participate in the study by the patient and/or parents or legal guardian after receipt of the study's information and non-objection note.

Ages: 11 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Left Ventricle Global Longitudinal 2D strain (LVGLS) expressed in percentage and obtained from cardiac ultrasound cineloop of 2D 4,3 and 2 apical views analyzed by the Tomtec STE Software. | 5 years
  To compare the evolution at 5 years ("Anthra2" study timeframe) of LVGLS obtained by STE analysis on patients treated with anthracyclines in childhood and previously included in first "Speckle Anthra" study, with the normal evolution of this parameter with age in healthy matched volunteers.

SECONDARY OUTCOMES:
Left Ventricle Ejection fraction (LVEF) by Simpson method (%) | The day of inclusion
  Compare the standard ultrasound parameter LVEF and the LVGLS obtained in "Speckle Anthra 2" on patients treated with anthracyclines in childhood and in the group of healthy volunteers.
Left ventricular myocardial dysfunction defined by LVEF < 55% | 5 years
  Correlation between the left ventricular myocardial dysfunction is defined by FeVG < 55% and the left global longitudinal 2D strain expressed in percentage and measured during the previous SpeckleAnthra study
Death secondary to toxic cardiomyopathy | 5 years
  Correlation between the rate of patients died with a toxic cardiomyopathy and the left global longitudinal 2D strain expressed in percentage and measured during the previous SpeckleAnthra study

OTHER OUTCOMES:
Known risk factors for cardiotoxicity | the day of inclusion
  To assess the effect of known risk factors for anthracycline cardiotoxicity, the anthracycline cumulative dose will be collected
Troponin T on the experimental group | The day of inclusion
  Troponin T is a biological markers of cardiotoxicity obtained in a standard blood test analysis and expressed in ng/ml. normal troponin value is between 0 and 0.04 ng/mL
NT-pro-BNP on the experimental group | The day of inclusion
  NT-pro-BNP (N terminal-pro-brain natriuretic peptides) is a biological markers of cardiotoxicity obtained in a standard blood test analysis and expressed in pg/ml. Normal NT-proBNP value is < 400pg/ml
Known risk factors for cardiotoxicity | the day of inclusion
  To assess the effect of known risk factors for anthracycline cardiotoxicity, young age at administration will be collected
Known risk factors for cardiotoxicity | the day of inclusion
  To assess the effect of known risk factors for anthracycline cardiotoxicity, female gender, will be collected
Known risk factors for cardiotoxicity | The day of inclusion
  To assess the effect of known risk factors for anthracycline cardiotoxicity, association with mediastinal radiotherapy will be collected

CONTACTS AND LOCATIONS:
Overall Officials: VINCENTI Marie, PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
sharing of results after obtaining
Supporting Information: Study Protocol, ICF
Time Frame: 5years
Access Criteria: Clinical trials
URL: https://clinicaltrials.gov

REFERENCES:
- [Background] Amedro P, Vincenti M, Abassi H, Lanot N, De La Villeon G, Guillaumont S, Gamon L, Mura T, Lopez-Perrin K, Haouy S, Sirvent A, Cazorla O, Vergely L, Lacampagne A, Avesani M, Sirvent N, Saumet L. Use of speckle tracking echocardiography to detect late anthracycline-induced cardiotoxicity in childhood cancer: A prospective controlled cross-sectional study. Int J Cardiol. 2022 May 1;354:75-83. doi: 10.1016/j.ijcard.2022.02.012. Epub 2022 Feb 12. PMID 35167907